CLINICAL TRIAL: NCT02211274
Title: Improving Veteran Transitions From VA Community Living Centers to the Community
Brief Title: VA Community Living Centers to Home
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to issues with the study, we did not proceed with enrolling participants in the trial.
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: D1241-W
Record Dates: First submitted 2014-07-31; First posted 2014-08-07 (Estimated); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Aged; Frail Elderly
Keywords: Quality of Life; Nursing Homes; Housing for the Elderly; Homes for the Aged

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study Group (Experimental): Individuals who want to leave the CLC will be allowed to participate in the study, there will be no assignment to groups. Individuals who want to leave the CLC will undergo transition care planning using the investigators' standardized toolkit. The investigators will compare outcomes to administrative data from other similar VA nursing homes.
  Interventions: Other: Everyday Competence Assessment and Planning for Community Transitions

INTERVENTIONS:
Other: Everyday Competence Assessment and Planning for Community Transitions — The Everyday Competence Assessment and Planning for Community Transitions (ECAP-CT) toolkit will allow CLC interdisciplinary team members to 1) assess the Veteran's everyday competence for safe and independent living; 2) develop personally meaningful rehabilitation goals that facilitate successful transition out of the CLC based on everyday competence; and 3) conduct structured treatment planning to support resident goals around transitioning back into the community. By considering everyday competence and goal-setting in this context, Veterans will have optimal P-E fit upon returning to the community, ensuring a successful transition.
  Other Names: ECAP - CT

SUMMARY:
Older adults prefer to live as in the community as long as possible. Creating a standardized treatment planning process that includes assessments of everyday competence and goal-setting techniques to help Veterans move from VA nursing homes back to the community can improve functional health, well-being, and quality of life for older Veterans. Research has shown that 29% of nursing home residents might be able to live safely in the community instead. Currently, VA provides nursing home care to more than 13,000 Veterans across the country, which costs about $3.3 billion a year. It is expensive for VA to provide nursing home care to these inappropriate residents and they are using limited resources that could be given to another Veteran with more urgent needs. The Everyday Competence Assessment and Planning for Community Transitions (ECAP-CT) toolkit will help these Veterans to move back into the community with the services and supports they need based on their individual level of everyday competence.

DETAILED DESCRIPTION:
Up to 29% of Community Living Center (CLC; VA nursing homes) residents may not require nursing home levels of care and could successfully reside in the community with appropriate rehabilitative services. Many older adults prefer to remain in their homes, though living independently in the community is not always possible or safe. According to the model of person-environment fit (P-E fit), older adults are at risk for poor outcomes when the demands and resources available in the living environment are not in balance with the individual's everyday competence (the ability to solve problems associated with everyday life). Community-dwelling older adults with low levels of everyday competence and little support are at risk for nursing home transition. Conversely, older adults with higher levels of everyday competence who live in more restrictive environments (e.g., nursing home) may experience declines in functioning resulting from a lack of stimulation. Often, transitions into nursing homes occur during a time of crisis (e.g., after acute hospital stay), leaving little opportunity for appropriate consideration of the individual's current and future level of everyday competence.

In VA, a major focus is to minimize the time spent in the CLCs by providing rehabilitation services and transitioning Veterans back into the community. The mission for the CLC program is to return the Veteran to his or her highest level of well-being, thus maximizing P-E fit. Despite this, CLC staff and Veterans face many barriers to facilitating transitions to the community (e.g., caregiving needs, housing, etc.). Currently no standardized process exists to assure that treatment planning includes processes to maximize P-E fit (e.g., assessing everyday competence, setting resident-directed goals around rehabilitation needs, and developing care plans to transition the Veteran to the community whenever possible).

The investigators' team has developed an instrument to allow providers to assess everyday competence for safe and independent living in the community. However, to ensure successful transitions, assessing everyday competence without intervention is not sufficient. Once CLC interdisciplinary team members have an understanding of the resident's everyday competence and barriers to transition, goal-setting must occur, focused on rehabilitation goals and care planning around transitioning to the community.

The objective of the proposed research is to develop an effective and feasible toolkit the CLC interdisciplinary team can use to 1) assess the Veteran's everyday competence for safe and independent living; 2) develop personally meaningful rehabilitation goals that facilitate successful transition out of the CLC based on everyday competence; and 3) conduct structured care planning to support resident goals around transitioning back into the community. With the innovative consideration of everyday competence and goal-setting in this context, Veterans will have optimal P-E fit upon returning to the community, thus ensuring a successful transition outcome (i.e., not readmitted to the CLC within 90 days).

ELIGIBILITY:
Inclusion Criteria:

* CLC residents will be included if they are able to demonstrate understanding of the informed consent process through teach-back and to communicate verbally.

Exclusion Criteria:

* CLC residents will be excluded if they are too cognitively impaired or have serious mental illness too severe to meaningfully participate in interviews (i.e., they are not "transition-capable").
* No participants will be excluded based on gender, race, social class, or ethnicity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Transition Outcome | 90 days post-discharge
  The primary outcome of interest for this pilot study will be transition outcome. Transitions will be "successful" if the resident leaves the CLC with a "community" destination and is not readmitted to the CLC within 90 days. For the purposes of this study, transitions to the "community" include any non-institutional environment that is more independent than the CLCs (e.g., single-family home, senior apartment, assisted living, medical foster home, etc.). For individuals who are unable to transition or who transition and are readmitted to the CLC within 90 days, these transitions will be "unsuccessful".

SECONDARY OUTCOMES:
Goal Attainment Scaling | Baseline
  An important outcome for participants at the intervention sites will be Goal Attainment Scaling64, which will allow us to identify if the resident was able to achieve the transition goals within the planned timeframe.
Multilevel Assessment Instrument - Environment Scale [MAI-ES] | Baseline and 90 days
  Measures person-environment fit
Multilevel Assessment Instrument - Environment Scale [MAI-ES] | 90 days
  Measures person-environment fit. Will be assessed at baseline and 90 days.
Multilevel Assessment Instrument - Environment Scale | Baseline and 90 days post discharge
  Measures person-environment fit.
Money Follows the Person - Quality of Life Scale | Baseline and 90 days post discharge
  Measures quality of life for individuals moving from a nursing home to the community.
Care Transitions Measure - 3 | Baseline and 90 days post discharge
  Measures individual's preparation for transitioning out of a health care facility.
Geriatric Depression Scale - Residential | Baseline and 90 days post discharge
  Measure of depression for older adults residing in residential care facilities.
Length of Stay in CLC | 30 days and 90 days post discharge
  Length of stay in the clc
Health Services Utilization | 30 days and 90 days post discharge
  Identify health services (e.g., hospital admission, ER visit, etc.) utilization following transition from CLC.

CONTACTS AND LOCATIONS:
Overall Officials: Whitney L. Mills, PhD, Principal Investigator — Providence VA Medical Center, Providence, RI
Locations (2):
- United States (2):
  - Providence VA Medical Center, Providence, RI, Providence, Rhode Island
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas

IPD SHARING:
Plan to Share IPD: No